CLINICAL TRIAL: NCT04991961
Title: Effect of Anti-hypertensive Medications on the Diagnostic Accuracy in Primary Aldosteronism：a Prospective Study
Brief Title: Effect of Anti-hypertensive Medications on the Diagnostic Accuracy in Primary Aldosteronism
Acronym: HASA
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Principal Investigator, Chongqing Medical University
Other Study IDs: HASA-China2020
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2020-09

CONDITIONS: Hypertension; Primary Aldosteronism
Keywords: hypertension; Aldosterone-Renin ratio; Primary aldosteronism
MeSH Terms: conditions — Hypertension; Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- primary aldosteronism group and essential hypertensin group: patients will be diagnosed as PA or EH based on ARR and CCT off interfering meds
  Interventions: Diagnostic Test: withdraw antihypertensive drugs
- primary aldosteronism (PA) group and essential hypertension (EH) group: The diagnosis of PA was established based on an ARR ≥20 pg·ml-1/μIU·ml-1 off interfering medications plus one of the following criteria: (1) PAC post-CCT off interfering medications was over 110pg/mL; (2) PAC post-CCT off interfering medications ranged from 80 to 110 pg/mL, but PAC post-SSIT off interfering medications exceeded 80 pg/mL. In patients with an ARR of 10-20 pg·ml-1/μIU·ml-1 but with hypokalemia or adrenal nodules, PA was also diagnosed if the confirmatory test was positive. The diagnosis of EH was determined if PA was excluded.
  Interventions: Diagnostic Test: withdraw antihypertensive drugs

INTERVENTIONS:
Diagnostic Test: withdraw antihypertensive drugs — patients need to withdraw of all antihypertensive drugs or change therapy to Doxazosin/Diltiazem for 2-4 weeks prior

SUMMARY:
To evaluate the effect of anti-hypertensive medication on efficiency of primary aldosteronism screening and confirmatory test, and to determine the appropriate diagnostic cutoff value for Chinese hypertension patients during antihypertensive drugs therapy.

DETAILED DESCRIPTION:
Aldosterone-Renin ratio (ARR)is currently the most reliable means available for screening for primary aldosterone（PA）while captopril challenging test is the widely used confirmatory test. However, some antihypertensive drugs may interfer aldosterone and renin levels. Thus, PA guidelines suggest that antihypertensive drugs should be withdraw or change therapy before screening.

But withdraw/changing the therapy is inconvenient for patients.

The investigators prepare to start a prospective study through recruiting hypertension patients, completing the ARR screening and captopril challenging test before and after withdraw/change therapy.

ELIGIBILITY:
Inclusion Criteria:

* Persistent hypertension >150/100mmHg, including previously diagnosed grade 2 hypertension but well controlled by 1-2 drugs; newly diagnosed hypertension with 3 days blood pressure > 150 / 100mmHg
* Resistant hypertension(combined with three antihypertensive drugs and one of them is diuretic but blood pressure is still greater than 140 / 90 mmHg ; or need to combined four anti-hypertensive drugs to control the blood pressure under 140 / 90 mmHg)
* Family history of hypertension with early onset (< 40 years old)
* Family history of hypertension with early onset (<40 years old) and cerebrovascular accident
* Hypertension with spontaneous or diuretic hypokalemia
* Hypertensive with adrenal incidentaloma
* Hypertensive with OSAS
* First-degree relatives of PA patients and with hypertension Stable antihypertensive medication therapy for more than 2 weeks, medication including：β-blockers, CCB, ACEi, ARB, MRA, and other diuretics.

Exclusion Criteria:

* Patients hard to change or stop the medication for accomplish the screening test or diagnosis Unwilling to participate the study and refuse to sign on informed consent Patients who was diagnosed with other secondary hypertension Suspected with PA（rein concretion beyond the limit of normal reference range after stoping or changing the medication） Severe renal insufficiency （eGFR<30 ml/min/1.73m2）; pregnancy

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the Department of Endocrinology and physical examination center of First Affiliated Hospital of CQMU who with hypertension, and under anti-hypertension medication therapy and being certificated with high risk factors of PA were recruited as the study group.
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Confirmation | 2 weeks
  Consistent diagnosis after drug withdrawal
Missing Diagnosis | 2 weeks
  essential hypertension turn to fit primary aldosteronism diagnosis after drug withdrawal
Misdiagnosis | 2 weeks
  primary aldosteronism turn to fit essential hypertension diagnosis after drug withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Li Qifu, PhD, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (2):
- China (2):
  - Qifu Li, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viola A, Monticone S, Burrello J, Buffolo F, Lucchiari M, Rabbia F, Williams TA, Veglio F, Mengozzi G, Mulatero P. Renin and aldosterone measurements in the management of arterial hypertension. Horm Metab Res. 2015 Jun;47(6):418-26. doi: 10.1055/s-0035-1548868. Epub 2015 May 8. PMID 25993253
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Schwartz GL, Turner ST. Screening for primary aldosteronism in essential hypertension: diagnostic accuracy of the ratio of plasma aldosterone concentration to plasma renin activity. Clin Chem. 2005 Feb;51(2):386-94. doi: 10.1373/clinchem.2004.041780. PMID 15681560
- [Background] Gallay BJ, Ahmad S, Xu L, Toivola B, Davidson RC. Screening for primary aldosteronism without discontinuing hypertensive medications: plasma aldosterone-renin ratio. Am J Kidney Dis. 2001 Apr;37(4):699-705. doi: 10.1016/s0272-6386(01)80117-7. PMID 11273868
- [Background] Niizuma S, Nakahama H, Kamide K, Fukuchi K, Iwanaga Y, Nakata H, Yoshihara F, Horio T, Nakamura S, Kawano Y. The cutoff value of aldosterone-to-renin ratio for the diagnosis of primary aldosteronism in patients taking antihypertensive medicine. Clin Exp Hypertens. 2008 Oct;30(7):640-7. doi: 10.1080/10641960802443282. PMID 18855267
- [Background] Young WF Jr. Diagnosis and treatment of primary aldosteronism: practical clinical perspectives. J Intern Med. 2019 Feb;285(2):126-148. doi: 10.1111/joim.12831. Epub 2018 Sep 25. PMID 30255616
- [Derived] Li X, Liang J, Hu J, Ma L, Yang J, Zhang A, Jing Y, Song Y, Yang Y, Feng Z, Du Z, Wang Y, Luo T, He W, Shu X, Yang S, Li Q; Chongqing Primary Aldosteronism Study (CONPASS) Group. Screening for primary aldosteronism on and off interfering medications. Endocrine. 2024 Jan;83(1):178-187. doi: 10.1007/s12020-023-03520-6. Epub 2023 Oct 5. PMID 37796417